CLINICAL TRIAL: NCT04500470
Title: Ketoprofen With or Without Vaginal Isonicotinic Acid Hydrazide (INH) Prior to Hysterosalpingography in Primarily Infertile Patients: a Randomized Controlled Trial
Brief Title: Ketoprofen With or Without Vaginal Isonicotinic Acid Hydrazide Prior to Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/351/3/19
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Ketoprofen; Isoniazid

STUDY DESIGN:
Intervention Model Description: double blind placebo randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind placebo randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): patients will have of oral Ketoprofen 60 minutes before the procedure plus 3 table 900 mg vaginal isonicotinic acid hydrazide by the patient 12 hours before the procedure
  Interventions: Drug: Ketoprofen + INH
- Group B (Placebo Comparator): patients will have of oral Ketoprofen 60 minutes before the procedure plus 3 table vaginal placebo by the patient 12 hours before the procedure
  Interventions: Drug: Ketoprofen + placebo

INTERVENTIONS:
Drug: Ketoprofen + INH — patients will have of oral Ketoprofen 60 minutes before the procedure plus 3 table 900 mg vaginal isonicotinic acid hydrazide by the patient 12 hours before the procedure
  Arms: Group A
Drug: Ketoprofen + placebo — patients will have of oral Ketoprofen 60 minutes before the procedure plus 3 table placebo by the patient 12 hours before the procedure
  Arms: Group B

SUMMARY:
The aim of our study is to determine the efficacy of Ketoprofen with or without vaginal isonicotinic acid hydrazide on the pain scores during HSG.

DETAILED DESCRIPTION:
hysterosalpingography can cause pain and discomfort in several ways: Use of the tenaculum to grasp the cervix and straighten the uterus for proper insertion; trans-cervical actions including measuring uterine depth, inserting the cannula; and injection of the dye

ELIGIBILITY:
Inclusion Criteria:

* any patient came for Hysterosalpingography

Exclusion Criteria:

* any patient has contraindication to HSG

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female candidate for 30 minutes after the procedure
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | 15 minutes
  pain during the procedure assessed by the visual analog scale from 0=no pain to 10 = the worst pain imaginable

SECONDARY OUTCOMES:
Intensity of pain | 30 minutes after the procedure
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure.visual analogue scale ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No